CLINICAL TRIAL: NCT05016635
Title: Disability-adjusted Life Years in a Senegalese Cohort of Patients With Subarachnoid Hemorrhage
Status: Completed | Type: Observational
Sponsor: Association of Future African Neurosurgeons, Yaounde, Cameroon (Other)
Responsible Party: Sponsor
Other Study IDs: AFANSEN1
Record Dates: First submitted 2021-08-17; First posted 2021-08-23 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Disability Adjusted Life Years of Sub-arachnoid Hemorrhage in Senegalese Cohort

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sub-arachnoid Hemorrhage Patients

SUMMARY:
Subarachnoid hemorrhage (SAH) is the extravasation of blood into the subarachnoid space from traumatic or nontraumatic origin. There is a paucity of data on the burden of SAH in African countries. In this study, we analyzed data from patients in the largest neurovascular center in Senegal to determine the sex- and age-adjusted burden of SAH in Senegal.

DETAILED DESCRIPTION:
The Fann Teaching Hospital (Dakar, Senegal) institutional review board authorized this study. Consent was obtained from adult patients and the parents/legal guardians of children. Patient data were stored in a password-protected Excel spreadsheet, and this spreadsheet was stored on a hard drive. Only the authors had access to the data.

ELIGIBILITY:
Inclusion Criteria:

* Sub-arachnoid Hemorrhage admission

Exclusion Criteria:

* Not admitted for sub-arachnoid hemorrhage

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We recruited 448 patients between 2011 and 2020. However, 60 patients (13.4%) had incomplete records and were excluded from the analysis. Herein we present the retrospective analysis of the 388 patients (86.6%) with complete records. We received a median of 40.0 patients annually (IQR=51.5), and a peak was observed in 2017 when 76 SAH patients were admitted at our institution.
Sampling Method: Probability Sample
Enrollment: 388 (Actual)
Dates: Start 2021-04-26 (Actual); Primary Completion 2021-08-16 (Actual); Study Completion 2021-08-16 (Actual)

PRIMARY OUTCOMES:
Disability Adjusted Life Years | 9 years
  Mortality and Morbidity

CONTACTS AND LOCATIONS:
Locations (1):
- Fann Teaching Hospital, Dakar, Senegal

IPD SHARING:
Plan to Share IPD: No